CLINICAL TRIAL: NCT07052201
Title: The Outcomes of Different Dexamethasone Regimens for the Prevention of Bronchopulmonary Dysplasia in Preterm Infants: A Multicenter Randomized Controlled Trial
Brief Title: Dexamethasone Regimens for BPD Prevention in Preterm Infants
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The Children's Hospital of Zhejiang University School of Medicine (Other)
Collaborators: Children's Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Yanping Xu, Principal Investigator, Department of NICU, The Children's Hospital of Zhejiang University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2025-IRB-0185-P-02
Record Dates: First submitted 2025-06-11; First posted 2025-07-04 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Infant, Premature; Bronchopulmonary Dysplasia (BPD)
MeSH Terms: conditions — Premature Birth; Bronchopulmonary Dysplasia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DART regimen (Experimental): DART regimen group (cumulative dose 0.89 mg/kg over 10 days)
  Interventions: Drug: Dexamethasone. Dart
- Medium-dose tapering regimen (Experimental): Medium-dose tapering regimen group (cumulative dose 2.35 mg/kg over 7 days)
  Interventions: Drug: Dexametasone. Medium

INTERVENTIONS:
Drug: Dexamethasone. Dart — DART regimen group (cumulative dose 0.89 mg/kg over 10 days): intravenous dexamethasone administered as follows:
  0.075 mg/kg/dose every 12 hours for 3 days 0.05 mg/kg/dose every 12 hours for 3 days 0.025 mg/kg/dose every 12 hours for 2 days 0.01 mg/kg/dose every 12 hours for 2 days, then discontinue.
  If extubation is not successful more than or equal to 2 weeks after completing the treatment, the regimen may be repeated.
  Arms: DART regimen
Drug: Dexametasone. Medium — Medium-dose tapering regimen group (cumulative dose 2.35 mg/kg over 7 days): intravenous dexamethasone administered as follows:
  0.5 mg/kg/d for 3 days 0.25 mg/kg/d for 3 days 0.1 mg/kg/d for 1 day If extubation is not successful more than or equal to 2 weeks after completing the treatment, the regimen may be repeated.
  Arms: Medium-dose tapering regimen

SUMMARY:
The goal of this clinical trial is to compare the effectiveness of two different dexamethasone treatment regimens (the DART regimen and the medium-dose tapering regimen) in reducing the incidence of Bronchopulmonary Dysplasia (BPD) or death by 36 weeks of postmenstrual age in premature infants. This study will also assess the safety of these treatments. The main questions it aims to answer are: Does the DART regimen, compared to the medium-dose tapering regimen, lower the rate of BPD or BPD-related death by 36 weeks of postmenstrual age in eligible premature infants? How do the two regimens compare in terms of short-term respiratory outcomes (like time to come off the ventilator), complications at hospital discharge, and long-term neurodevelopmental outcomes at 18-24 months of corrected age?

Researchers will compare the DART regimen group (lower cumulative dose, given over 10 days) to the medium-dose tapering regimen group (higher cumulative dose, given over 7 days) to see which one is more effective and safer.

Participants will:

Inclusion Criteria (Must meet ALL of the following)

1. Gestational age 24+0 to 29+6 weeks; requires invasive mechanical ventilation for ≥14 days after birth; within 14-28 days of age at first receive of dexamethasone.
2. FiO₂ > 40% and MAP > 8 cmH₂O (maintained for at least 24 hours prior to enrollment).
3. Parent/Legal guardian has provided signed informed consent.
4. No use of other steroid medications prior to enrollment, as explicitly stated in the inclusion criteria.

2. Exclusion Criteria (Will be excluded if they meet ANY of the following)

1. Presence of ventilator-associated pneumonia at the time of enrollment.
2. Severe congenital malformations (e.g., severe cardiac anomalies, congenital diaphragmatic hernia, etc.), or known immunodeficiency.
3. Suffering from other severe life-threatening illnesses with a short-expected survival time.
4. Parent/Legal guardian refuses to participate in the study.

DETAILED DESCRIPTION:
This study is a multicenter, prospective, randomized, parallel-controlled clinical trial.

Study Sites: Multiple hospitals across China with high-level Neonatal Intensive Care Units (NICUs) will participate.

Randomization:

A randomization method will be used to assign participants to one of two study groups in a 1:1 ratio. Subjects will receive a unique randomization number in the order of enrollment and will be assigned to one of the following treatment groups:

* DART regimen
* Moderate-dose tapering regimen

Blinding:

Blinding will be applied for the assessment of secondary outcomes (e.g., neurodevelopmental outcomes). Evaluators will be from an independent team and will not be involved in the routine clinical care of the infants.

1. DART Regimen Group

   Cumulative dose: 0.89 mg/kg over 10 days Intravenous dexamethasone [17], administered as follows:
   * 0.075 mg/kg/dose, every 12 hours for 3 days
   * 0.05 mg/kg/dose, every 12 hours for 3 days
   * 0.025 mg/kg/dose, every 12 hours for 2 days
   * 0.01 mg/kg/dose, every 12 hours for 2 days, then discontinue

   If extubation is not successful more than or equal to two weeks after completing the treatment (FiO2 > 40% and MAP > 8 cmH2O), the DART regimen may be repeated. The number of repeated courses, reasons, and specific timing must be documented.

   (Note: According to reference [13], if the infant meets respiratory criteria again at least 72 hours after completing the initial 9-day course, a second 9-day course may be administered. If the infant meets the criteria again during the 42-day observation period, a third course may be considered.)

   Rationale for design:

   Due to the rapid physiological changes in preterm infants, early responses to interventions are often evident within short timeframes. The shorter assessment intervals aim to capture early treatment effects more sensitively and dynamically.

   Previous exploratory observations indicated that two-week intervals are feasible and safe for evaluating parameters such as weight gain and lab changes, with no significant adverse effects observed.
2. Moderate-Dose Tapering Regimen Group

Cumulative dose: 2.35 mg/kg over 7 days Intravenous dexamethasone [19], administered as follows:

* 0.5 mg/kg/d for 3 days
* 0.25 mg/kg/d for 3 days
* 0.1 mg/kg/d for 1 day

If extubation is not successful more than or equal to two weeks after completing the treatment (FiO2 > 40% and MAP > 8 cmH2O), the same regimen may be repeated. The number of repeated courses, reasons, and specific timing must be documented.

Definition of BPD Severity (based on 2019 consensus criteria):

Clinically, BPD is defined as oxygen and/or respiratory support dependency for at least 28 days or continuing until 36 weeks corrected gestational age in preterm infants born at <32 weeks gestation.

ELIGIBILITY:
Inclusion Criteria (Must meet ALL of the following)

1. Gestational age 24+0 to 29+6 weeks; requires invasive mechanical ventilation for ≥14 days after birth; within 14-28 days of age at first receive of dexamethasone.
2. FiO₂ > 40% and MAP > 8 cmH₂O (maintained for at least 24 hours prior to enrollment).
3. Parent/Legal guardian has provided signed informed consent.
4. No use of other steroid medications prior to enrollment, as explicitly stated in the inclusion criteria.

Exclusion Criteria (Will be excluded if they meet ANY of the following)

1. Presence of ventilator-associated pneumonia at the time of enrollment.
2. Severe congenital malformations (e.g., severe cardiac anomalies, congenital diaphragmatic hernia, etc.), or known immunodeficiency.
3. Suffering from other severe life-threatening illnesses with a short-expected survival time.
4. Parent/Legal guardian refuses to participate in the study.

Ages: 14 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 970 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Bronchopulmonary dysplasia (BPD) and/or death at 36 weeks corrected age | 36 weeks PMA
  Two different dexamethasone treatment regimens (DART regimen and moderate-dose tapering regimen) on the incidence of Bronchopulmonary dysplasia (BPD) and/or death at 36 weeks corrected age in preterm infants meeting inclusion criteria
  BPD severity will be assessed at 36 weeks postmenstrual age (PMA) using the Jensen Criteria for BPD Severity, a categorical classification system. The Jensen Criteria define BPD severity based on the mode of respiratory support required at 36 weeks PMA:
  Grade 0: No BPD (no respiratory support) Grade 1: Nasal cannula ≤2 L/min Grade 2: Nasal cannula >2 L/min or non-invasive positive airway pressure (e.g., continuous positive airway pressure (CPAP)), or noninvasive intermittent positive pressure ventilation (NIPPV) Grade 3: Invasive mechanical ventilation Higher grades represent worse outcomes (i.e., more severe BPD).

SECONDARY OUTCOMES:
Extubation Rate (72 hours) | 72 hours
  Weaning from the ventilator for more than 72 hours after the first course of dexamethasone
Extubation Rate (7 days) | 7 days
  Weaning from the ventilator for more than 7 days after the first course of dexamethasone.
Incidence of Adverse Events Including Intestinal Perforation, Hyperglycemia, Hypertension, Infection, and Gastrointestinal Bleeding Following Dexamethasone Administration | Within 72 hours and 7 days after dexamethasone administration
  Assessment of the number and type of adverse events related to dexamethasone administration, specifically monitoring for intestinal perforation, hyperglycemia, hypertension, infection, and gastrointestinal bleeding.
Oxygenation index | Baseline (Day 0) and on Days 3, 7, 10, 14, 28 Following Dexamethasone Therapy
  OI= (MAP × FiO₂ ×100 / PaO₂)
Total Duration of Invasive Mechanical Ventilation During Initial Hospitalization | From birth until hospital discharge (up to approximately 44 weeks postmenstrual age)
  This outcome measures the cumulative number of days each participant receives invasive mechanical ventilation (via endotracheal tube) during the initial hospitalization from birth until discharge. This includes all consecutive and non-consecutive days on invasive respiratory support. The data will be reported in days.
Total Length of Initial Hospitalization (Days from Birth to Discharge) | From birth until hospital discharge (up to approximately 44 weeks postmenstrual age )
  This outcome measures the total number of days each participant remains hospitalized from birth until initial hospital discharge. The duration is counted in calendar days, including any days spent in transfer between hospitals if part of the initial hospitalization period. The expected maximum timeframe is up to approximately 44 weeks PMA, depending on gestational age at birth.
Incidence of Neonatal Complications Including ROP, IVH, Hemodynamically Significant PDA, Late-Onset Sepsis, PVL, NEC, SIP, Short Bowel Syndrome, and Pulmonary Hypertension | From birth until hospital discharge (up to approximately 44 weeks postmenstrual age)
  This measure will capture the incidence of various neonatal complications occurring from birth until the time of hospital discharge. Complications include:
  Retinopathy of Prematurity (ROP) Intraventricular Hemorrhage (IVH) Hemodynamically Significant Patent Ductus Arteriosus (HsPDA) Late-Onset Sepsis Periventricular Leukomalacia (PVL) Necrotizing Enterocolitis (NEC) Spontaneous Intestinal Perforation (SIP) Short Bowel Syndrome Pulmonary Hypertension Each diagnosis is based on clinical evaluation and/or standardized diagnostic criteria during the neonatal hospitalization period. The maximum follow-up duration is expected to be approximately 44 weeks PMA.
Bayley Scales of Infant and Toddler Development, Third Edition (Bayley-III) - Cognitive Composite Score (MDI) | At 18 to 24 months corrected age
  The Bayley-III Cognitive Composite Score (formerly referred to as the Mental Development Index, MDI) assesses cognitive development.
  Score Range: 55 (minimum) to 145 (maximum) Mean: 100 Standard Deviation: 15 Interpretation: Higher scores indicate better cognitive outcomes.
Bayley Scales of Infant and Toddler Development, Third Edition (Bayley-III) - Motor Composite Score (PDI) | At 18 to 24 months corrected age
  The Bayley-III Motor Composite Score (formerly referred to as the Psychomotor Development Index, PDI) assesses fine and gross motor development.
  Score range: 55 (minimum) to 145 (maximum) Mean: 100, Standard Deviation: 15 Higher scores indicate better motor outcomes
Griffiths Mental Development Scales - General Development Score | At 18 to 24 months corrected age
  The Griffiths Mental Development Scales assess multiple developmental domains in infants and toddlers.
  Score range: Typically 50 to 150 (depending on version) Mean: 100, Standard Deviation: 15 Higher scores indicate better developmental outcomes

CONTACTS AND LOCATIONS:
Locations (24):
- China (24):
  - Children's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Chengdu Maternal and Children's Health Care Hospital, Chengdu
  - Children's Hospital of Chongqing Medical University, Chongqing
  - Women and Children's Hospital of Chongqing Medical University, Chongqing
  - Guangdong Women and Children Hospital, Guangdong
  - Guangxi Maternal and Child Health Hospital, Guangxi
  - Guiyang Maternity and Child Health Care Hospital, Guiyang
  - Guizhou Provincial People's Hospital, Guizhou
  - The First Hospital of Jilin University, Jilin
  - First Affiliated Hospital of Kunming Medical University, Kunming
  - Jiangxi Maternal and Child Health Hospital, Nanchang
  - Nanjing Maternity and Child Health Care Hospital, Nanjing
  - Ningbo Women & Children's Hospital, Ningbo
  - QuanZhou Women and Children's Hospital, Quanzhou
  - Qujing Maternal and Child Health Hospital, Qujing
  - Shanghai Children's Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai
  - Xinhua Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai
  - Shengjing Hospital, Shengyang
  - Shenzhen Maternal and Child Health Hospital, Shenzhen
  - Fourth Hospital of Shijiazhuang City, Shijiazhuang
  - Xiamen Women's and Children's Hospital, Xiamen
  - First Affiliated Hospital of Xinjiang Medical University, Xinjiang
  - Zhangzhou Affiliated Hospital of Fujian Medical University, Zhangzhou
  - Zhengzhou Children's Hospital, China, Zhengzhou

IPD SHARING:
Plan to Share IPD: Undecided
After the article was published

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-09-26): https://cdn.clinicaltrials.gov/large-docs/01/NCT07052201/Prot_SAP_ICF_002.pdf